CLINICAL TRIAL: NCT06236451
Title: A Randomized Controlled Trial to Evaluate Atypical Antipsychotic-induced Mitochondrial Dysfunction in Patients With Schizophrenia
Brief Title: Atypical Antipsychotic-induced Mitochondrial Dysfunction in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGThesis/2023-24/100
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mitochondrial electron transport chain complex; Aripiprazole; Risperidone; Mitochondrial dysfunction
MeSH Terms: conditions — Schizophrenia; Mitochondrial Diseases | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole group (Experimental): Aripiprazole will be started at dose of 10 mg/day and increased to a stable dose of 20 mg/day over 2-3 weeks and will be continued till 12 weeks.
  Interventions: Drug: Aripiprazole
- Risperidone group (Active Comparator): Risperidone will be started at dose of 2 mg/day and increased to a stable dose of 6 mg/day over 2-3 weeks and continued till 12 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole will be started at dose of 10 mg/day and increased to a stable dose of 20 mg/day over 2-3 weeks and will be continued till 12 weeks.
  Arms: Aripiprazole group
Drug: Risperidone — Risperidone will be started at dose of 2 mg/day and increased to a stable dose of 6 mg/day over 2-3 weeks and continued till 12 weeks.
  Arms: Risperidone group

SUMMARY:
Schizophrenia is a serious mental disorder with a global prevalence of 1%. The main cause of this condition is dysfunction in the signaling of neurotransmitters dopamine, serotonin, glutamate and Gamma-aminobutyric acid .According to recent research, a disturbed cellular energy state caused by mitochondrial dysfunction is thought to be a factor in the development of schizophrenia.

The aim of the treatment of schizophrenia is to reduce symptoms and is mainly based on the monoamine hypothesis. Atypical antipsychotics are the first-line of treatment.

Certain typical and atypical antipsychotic medications have been shown in prior preclinical research to decrease mitochondrial respiratory chain complex I activity. In contrast to individuals who were drug-naive, Casademont et al. found a significant decrease in complex I activity with haloperidol and risperidone in one cross-sectional observational study. Also, there is evidence suggesting that mitochondrial dysfunction is linked to the extrapyramidal side effects seen with antipsychotics.

To date, there are no randomized controlled trials that assess the effect of these drugs on mitochondrial functions. Hence, the present randomized controlled trial has been planned to evaluate and compare the clinical and biochemical markers of mitochondrial dysfunction in schizophrenia patients treated with the atypical antipsychotics risperidone and aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the DSM-5 criteria for diagnosis of schizophrenia.
* Treatment naıv̈ e patients or patients who had not taken any antipsychotic drugs for at least 4 weeks before recruitment.
* Patients of either sex between the ages of 18 and 60 years.
* Legally authorized representative (LAR) of patients consenting to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Patients diagnosed with other psychiatric disorders including schizoaffective disorder or schizophrenia with somatoform disorders.
* Highly agitated patients who need immediate indoor-based treatment.
* Patients with known mitochondrial disorders (MELAS, LHON, Leigh syndrome, KearnsSayre syndrome, MERRF etc.)
* Patients with history of comorbidities like cardiovascular, renal, hepatic, neurological, respiratory or endocrinal diseases or malignancies.
* Patients with history of substance abuse.
* Pregnant or lactating mothers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Change in Mitochondrial respiratory chain complex I activity/concentration | 12 weeks
  Mitochondrial respiratory chain complex I activity/concentration will be measured in platelets using a commercially available ELISA (enzyme-linked immunosorbent assay) kit at baseline and at 12 weeks of follow-up.

SECONDARY OUTCOMES:
Change in Serum lactate | 12 weeks
  Serum lactate will be measured using spectrophotometry at baseline and at 12 weeks follow up
Change in Serum creatine kinase | 12 weeks
  Serum creatine kinase will be measured using autoanalyzer at baseline and at 12 weeks
Change in Newcastle Mitochondrial Disease Adult Scale (NMDAS) scores | 12 weeks
  Newcastle Mitochondrial Disease Adult Scale (NMDAS) scoring of all patients will be assessed at baseline and at 12 weeks of follow-up. The NMDAS offers a range of 0 to 5 points for each question. The results from each of the first three sections' questions are added together to determine each section's score. The more severe the ailment, the higher the score.
Change in Positive and Negative Syndrome Scale (PANSS) scores | 12 weeks
  Positive and Negative Syndrome Scale (PANSS) scoring will be done at baseline and at 12 weeks follow-up. Out of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale. The scores for these scales are arrived at by summation of ratings across component items. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. The more severe the ailment, the higher the score.
Responder rate | 12 weeks
  A patient with a reduction of Positive and Negative Syndrome Scale (PANSS) scores by ≥50% from baseline will be considered a 'responder'..
Change in Serum pyruvate | 12 weeks
  Serum pyruvate will be measured using spectrophotometry at baseline and at 12 weeks follow up.
Incidence of treatment-emergent adverse events | 12 weeks
  Incidence of treatment-emergent adverse events in both study groups reported throughout the study duration will be reported.
Severity of extrapyramidal adverse effects | 12 weeks
  Total score severity of extrapyramidal adverse effects will be assessed by Modified Simpson-Angus Scale. It is a 10-item scale where each item is rated on a 0-4 scale, with higher scores indicating greater severity. The total score is used to gauge the presence and degree of movement disorders, ranging from normal (score<3) to severe (score>12).

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this study will be shared with qualified researchers upon reasonable request. Data will be available after publication and subject to review of a data access proposal and data use agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after publication and will be available for 5 years after publication.
Access Criteria: Data will be shared with qualified researchers upon reasonable request and subject to review of a data access proposal and data use agreement.

REFERENCES:
- [Result] Hardy RE, Chung I, Yu Y, Loh SHY, Morone N, Soleilhavoup C, Travaglio M, Serreli R, Panman L, Cain K, Hirst J, Martins LM, MacFarlane M, Pryde KR. The antipsychotic medications aripiprazole, brexpiprazole and cariprazine are off-target respiratory chain complex I inhibitors. Biol Direct. 2023 Aug 1;18(1):43. doi: 10.1186/s13062-023-00375-9. PMID 37528429
- [Result] Luptak M, Fisar Z, Hroudova J. Effect of Novel Antipsychotics on Energy Metabolism - In Vitro Study in Pig Brain Mitochondria. Mol Neurobiol. 2021 Nov;58(11):5548-5563. doi: 10.1007/s12035-021-02498-4. Epub 2021 Aug 8. PMID 34365585
- [Result] Modica-Napolitano JS, Lagace CJ, Brennan WA, Aprille JR. Differential effects of typical and atypical neuroleptics on mitochondrial function in vitro. Arch Pharm Res. 2003 Nov;26(11):951-9. doi: 10.1007/BF02980205. PMID 14661862
- [Result] Scaini G, Rochi N, Morais MO, Maggi DD, De-Nes BT, Quevedo J, Streck EL. In vitro effect of antipsychotics on brain energy metabolism parameters in the brain of rats. Acta Neuropsychiatr. 2013 Feb;25(1):18-26. doi: 10.1111/j.1601-5215.2012.00650.x. PMID 26953070
- [Result] Casademont J, Garrabou G, Miro O, Lopez S, Pons A, Bernardo M, Cardellach F. Neuroleptic treatment effect on mitochondrial electron transport chain: peripheral blood mononuclear cells analysis in psychotic patients. J Clin Psychopharmacol. 2007 Jun;27(3):284-8. doi: 10.1097/JCP.0b013e318054753e. PMID 17502776
- [Result] Rajasekaran A, Venkatasubramanian G, Berk M, Debnath M. Mitochondrial dysfunction in schizophrenia: pathways, mechanisms and implications. Neurosci Biobehav Rev. 2015 Jan;48:10-21. doi: 10.1016/j.neubiorev.2014.11.005. Epub 2014 Nov 15. PMID 25446950
- [Result] Fizikova I, Dragasek J, Racay P. Mitochondrial Dysfunction, Altered Mitochondrial Oxygen, and Energy Metabolism Associated with the Pathogenesis of Schizophrenia. Int J Mol Sci. 2023 Apr 28;24(9):7991. doi: 10.3390/ijms24097991. PMID 37175697
- [Result] Schaefer AM, Phoenix C, Elson JL, McFarland R, Chinnery PF, Turnbull DM. Mitochondrial disease in adults: a scale to monitor progression and treatment. Neurology. 2006 Jun 27;66(12):1932-4. doi: 10.1212/01.wnl.0000219759.72195.41. PMID 16801664
- [Result] Leucht S, Davis JM, Engel RR, Kane JM, Wagenpfeil S. Defining 'response' in antipsychotic drug trials: recommendations for the use of scale-derived cutoffs. Neuropsychopharmacology. 2007 Sep;32(9):1903-10. doi: 10.1038/sj.npp.1301325. Epub 2007 Feb 7. PMID 17287825
- [Result] Venegas V, Halberg MC. Measurement of mitochondrial DNA copy number. Methods Mol Biol. 2012;837:327-35. doi: 10.1007/978-1-61779-504-6_22. PMID 22215558
- [Derived] Shaju A, Mohapatra D, Mishra BR, Mishra A, Srinivasan A, Maiti R. Evaluation of atypical antipsychotic-induced mitochondrial dysfunction in patients with schizophrenia: a randomised controlled trial protocol. BMJ Open. 2025 Oct 15;15(10):e098173. doi: 10.1136/bmjopen-2024-098173. PMID 41093357